CLINICAL TRIAL: NCT05017883
Title: TAA05 Cell Injection in the Treatment of Recurrent / Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V2.0
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-08

CONDITIONS: CAR; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAA05 cell injection (Experimental): TAA6 cell injection#Targeting FLT3 autologous chimeric antigen receptor T cells#
  Interventions: Drug: TAA05 cell injection

INTERVENTIONS:
Drug: TAA05 cell injection — Chimeric antigen receptor T cells (car-t)
  Chimeric antigen receptor T cells (car-t) is one of the most effective therapies for malignant tumors (especially hematological tumors). Like other immunotherapies, the basic principle is to use the patient's own immune cells to clear cancer cells. Chimeric antigen receptor (car) is the core component of car-t, which endows T cells with the ability to recognize tumor antigens in an independent manner,which enables car modified T cells to recognize a wider range of targets than natural T cell surface receptors (TCR). The basic design of car includes a tumor associated antigen binding region (usually derived from scFv segment of monoclonal antibody antigen binding region), transmembrane region and intracellular signal region. The selection of target antigen is a key determinant for the specificity and effectiveness of car and the safety of genetically modified T cells.

SUMMARY:
This is a clinical study of ytaa05 cell injection in the treatment of patients with recurrent / refractory acute myeloid leukemia.The purpose is to evaluate the safety and preliminary efficacy of FLT3 car-t cells in patients with recurrent / refractory FLT3 positive acute myeloid leukemia.#TAA05 cell injection is a T cell targeting FLT3 chimeric antigen receptor#

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a hematological malignancy caused by abnormal differentiation and uncontrolled proliferation of hematopoietic progenitor cells. If AML is not given active treatment within one year after diagnosis, it will cause fatal infection, bleeding and organ infiltration due to abnormal proliferation of tumor cells. AML is one of the most common leukemia. About 3.8 patients in every 100000 people are in the higher incidence rate among people aged 65 and over, and 17.9 patients in every 100000 people. The cure rate of AML is about 35-40% in patients ≤ 60 years old and only 5-15% in patients over 60 years old. The survival of elderly patients who can not tolerate chemotherapy is frustrating, and the median survival time is only 5-10 months. In the past 20 to 30 years, the treatment of acute myeloid leukemia (AML) has made significant progress, so that about 80% of adult patients under the age of 55 can achieve complete remission. However, more than half of Cr patients will relapse, and the long-term survival rate is about 40%. Until the 1970s, diagnosis was only based on pathological and cytological examination of bone marrow and blood. The five-year survival rate was less than 15%.

CAR-T cells can recognize specific antigens in a non restricted manner of HLA and continuously activate T cells. FLT3 is a potential target of AML. Therefore, the construction of car-t cells that recognize human FLT3 molecule has high clinical value in the treatment of AML.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 70 years old (including boundary value), regardless of gender;
2. Acute myeloid leukemia with FLT3 positive (positive rate ≥ 30%) verified by flow cytometry or immunohistochemistry;
3. The expected survival time was more than 12 weeks;
4. ECoG score 0-2;
5. Refractory or relapse after standardized treatment;
6. Liver and kidney function and cardiopulmonary function meet the following requirements:

   1. Creatinine ≤ 1.5 ULN;
   2. Left ventricular ejection fraction ≥ 45%;
   3. Blood oxygen saturation > 91%;
   4. Total bilirubin ≤ 1.5 × ULN； ALT and AST ≤ 2.5 × ULN；
7. Understand the test and have signed the informed consent form.

Exclusion Criteria:

1. Patients with graft-versus-host disease (GVHD) or requiring immunosuppressive agents;
2. Malignant tumors other than acute myeloid leukemia within 5 years before screening, except fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical operation, and breast ductal carcinoma in situ after radical operation;
3. hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal reference range; Hepatitis C virus (HCV) antibody positive and hepatitis C virus (HCV) RNA positive in peripheral blood; Human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA positive; Syphilis test positive;
4. Severe heart disease: including but not limited to unstable angina pectoris, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade III), severe arrhythmia;
5. Unstable systemic diseases judged by the researcher: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
6. Within 7 days before screening, there were active or uncontrollable infections requiring systemic treatment (except mild urogenital infection and upper respiratory tract infection);
7. Pregnant or lactating women, female subjects who planned pregnancy within 1 year after cell reinfusion, or male subjects whose partners planned pregnancy within 1 year after cell reinfusion;
8. Those who had received car-t therapy or other gene modified cell therapy before screening;
9. Subjects who were receiving systemic steroid treatment within 7 days before screening or who were determined by the investigator to need long-term systemic steroid treatment during treatment (except inhalation or local use);
10. Participated in other clinical studies within 3 months before screening;
11. There was evidence of central nervous system invasion during subject screening;
12. According to the judgment of the researcher, it does not conform to the situation of cell preparation;
13. Other researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
ORR 3 ORR 3 | three months after CAR-T cells infusion
  3-month objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Xingbing Wang, Principal Investigator — No.1, Swan Lake Road, new administrative and Cultural District, Hefei City, Anhui Province
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China